CLINICAL TRIAL: NCT04572152
Title: A Phase 1a/1b, Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, and Anti-tumor Activity of AK119 in Combination With AK104 in Subjects With Advanced or Metastatic Solid Tumors.
Brief Title: A Study of AK119 (Anti-CD73) in Combination With AK104 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK119-102
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Anti CD73; PD-1/ CTLA-4; Bispecific

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK119/ AK104 (Experimental): Single-arm
  Interventions: Biological: AK119; Biological: AK104

INTERVENTIONS:
Biological: AK119 — Subjects will receive AK119 by intravenous administration.
Biological: AK104 — On the same day subjects will receive AK104 by intravenous administration.

SUMMARY:
This is a first-in-human (FIH), Phase 1a/1b, Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, and Anti-tumor Activity of AK119 (Anti-CD73) in Combination with AK104 in Subjects with Advanced or Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Age ≥ 18 years.
3. In dose-escalation cohorts (Phase 1a), subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor that is refractory or relapsed to the current standard therapies, or for which no effective standard therapy is available, or whereby standard therapy has been refused.
4. In pharmacodynamic-confirmation cohorts (Phase 1a), additional enrolled subjects must have histologically or cytologically confirmed selected advanced or metastatic solid tumors, refractory or relapsed to the current standard therapies, or for which no effective standard therapy is available. Other tumor types can be considered after discussion with the Sponsor.
5. In dose-expansion cohorts (Phase 1b), subjects with specific tumor types will be enrolled. Subjects must have received no more than three prior lines of systemic therapy (including approved and investigational treatments) for advanced or metastatic disease. Other cohorts of different tumor types may be added based on the emerging pharmacodynamic and anti-tumor response data.
6. Subjects must have measurable lesions according to RECIST v1.1. A previously irradiated lesion can be considered a target lesion if the lesion is measurable per RECIST v1.1, and there is objective evidence of interval increase in size since radiotherapy.
7. For dose-escalation cohorts (Phase 1a), subjects must have available archived tumor tissue sample (block or a minimum of 10 unstained slides of formalin-fixed paraffin-embedded [FFPE] tissues) to allow for correlative biomarker studies.
8. For pharmacodynamic-confirmation cohorts (Phase 1a) and dose-expansion cohorts (Phase 1b), subjects must be willing to provide 2 fresh biopsy samples (pre-treatment and on treatment), where clinically appropriate.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to1.
10. Adequate organ function
11. Life expectancy ≥12 weeks;
12. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and within 120 days after the last dose of investigational product.
13. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and within 120 days after the last dose of investigational product.

Exclusion Criteria:

1. Receipt of the following treatments or procedures:

   1. Anticancer small-molecule targeted agent (e.g., tyrosine kinase inhibitor) within 2 weeks prior to the first dose of investigational product;
   2. Anti-PD-1/PD-L1 mAb within 4 weeks prior to the first dose of investigational product;
   3. Prior use of approved or investigational anti-CTLA-4 therapy, anti-CD73 therapy or adenosine 2A receptor inhibitors, or any other antibody or drug targeting T cell costimulation or immune checkpoint pathways such as ICOS, or agonists such as CD40, CD137, GITR, OX40 etc.
   4. Other anticancer mAb within 4 weeks or 5 half-lives (whichever is less) prior to the first dose of investigational product;
   5. Other anticancer therapy (e.g., chemotherapy, radiotherapy, etc.) within 4 weeks prior to the first dose of investigational product; [Note: Palliative radiotherapy > 1 week prior to first dose is allowed]
   6. Any major surgery (e.g., laparotomy, thoracotomy, removal of organ[s]) within 4 weeks prior to the first dose of investigational product;
   7. Any other non-approved investigational product or procedure within 4 weeks prior to the first dose of investigational product, or concurrent participation in another therapeutic clinical study;
2. Any condition that required systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of investigational product.
3. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of investigational product; Note: seasonal vaccine for influenza which is generally inactivated is allowed.
4. Prior organ transplantation;
5. Prior malignancy active within the previous 3 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured, such as basal cell cancer or carcinoma in situ of the cervix or breast;
6. Subjects with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at Screening (based on 2 sets of brain images, performed ≥ 4 weeks apart, and obtained after the brain metastases treatment).
7. Active infections (including tuberculosis) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to the first dose of investigational products. Note: antiviral therapy is permitted for patients with viral hepatitis;
8. Known history of human immunodeficiency virus (HIV) infection;
9. Known active hepatitis B or C infections (Active hepatitis B is defined as a known positive Hepatitis B surface antigen [HBsAg] result. Active hepatitis C is defined by a known positive Hepatitis C virus [HCV] antibody with detectable HCV ribonucleic acid [RNA] results);
10. Active autoimmune diseases or history of autoimmune diseases that may relapse. Note: Subjects with controlled type 1 diabetes mellitus, thyroiditis in euthyroid state or hypothyroidism well managed by hormone replacement therapy (HRT), or skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis) are eligible;
11. History of interstitial lung disease, noninfectious pneumonitis except for those induced by radiation therapies;
12. Uncontrolled massive ascites or pleural effusion, as determined by the Investigator;
13. Patients with clinically significant cardio-cerebrovascular or venous thromboembolic disease.
14. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec calculated from 3 ECGs (within 5 minutes at least 1 minute apart);
15. Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, uncontrolled diabetes, uncontrolled endocrinopathy, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent;
16. History of severe hypersensitivity reactions to other mAbs;
17. Toxicities of prior anticancer therapy have not resolved to NCI-CTCAE version 5.0 Grade ≤1, or to levels dictated in the inclusion/exclusion criteria, except toxicities not considered a safety risk (e.g., alopecia, neuropathy, or asymptomatic laboratory abnormalities);
18. Pregnant or breastfeeding women;
19. Any other conditions that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 6 weeks
  DLTs will be assessed during the first 6 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 6 weeks of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Maximum observed concentration (Cmax) of AK119 and AK104 | From first dose of study drug through 30 days after last dose of study drug
  The endpoints for assessment of PK include serum concentrations of AK119 and AK104 at different timepoints after study drug administration.
Minimum observed concentration (Cmin) of AK119 and AK104 at steady state | From first dose of study drug through 30 days after last dose of study drug
  The endpoints for assessment of PK include serum concentrations of AK119 and AK104 at different timepoints after study drug administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 90 days after last dose of study drug
  The immunogenicity of AK119 and AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Blacktown Cancer and Haematology Centre (Blacktown Hospital), Blacktown, New South Wales
  - ICON Cancer Centre, South Brisbane, Queensland
  - Ashford Cancer Centre, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Alfred Health (The Alfred Hospital), Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No